CLINICAL TRIAL: NCT06019923
Title: Study on the Dynamic Changes of Metabolic Biomarkers and Their Prognostic Relationship in Ovarian Cancer
Status: Recruiting | Type: Observational
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB-20230265-R
Record Dates: First submitted 2023-08-24; First posted 2023-08-31 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The collected plasma samples are used for plasma metabolomics analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Ovarian cancer is a highly lethal gynecological malignancy, often diagnosed at an advanced stage, with high rates of recurrence within 1-2 years after frontline treatment. Current guidelines recommend monitoring tumor markers CA125 and HE4 for disease progression, but these markers may not detect recurrence or disease progression when their levels are below the detection limit. Therefore, there is a need to identify new prognostic biomarkers and monitor their dynamic changes for effective risk stratification and personalized treatment in patients with ovarian cancer

DETAILED DESCRIPTION:
Ovarian Cancer is the deadliest gynecological malignancy, with over 70% of patients being diagnosed at advanced stages, and more than 70% experiencing recurrence within 1-2 years after frontline treatment. The recommended tumor biomarkers for monitoring ovarian cancer progression, CA125 and HE4, still pose the risk of recurrence and disease progression when their levels are below the detection limit. Therefore, it is of paramount importance to search for new prognostic monitoring biomarkers for ovarian cancer in order to stratify the prognosis and implement personalized treatment, ultimately improving patient outcomes. Previous research and literature have indicated that metabolic biomarkers can directly reflect the biochemical changes, physiological status, and disease progression in cancer patients. In comparison to studying the relationship between metabolite expression levels at a single time point and disease prognosis, the dynamic changes in metabolite trajectories with multiple time points can better reflect the dynamic patterns of disease progression throughout the entire cancer cycle, providing more prognostic information for patients with ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years;
* Pathological diagnosis of high-grade serous ovarian cancer;
* Newly diagnosed ovarian cancer case without prior neoadjuvant therapy.

Exclusion Criteria:

* Non-primary (recurrent) patients;
* Ovarian cancer patients who have not undergone surgical treatment;
* Patients with a history of other malignancies.

Ages: 18 Years to 75 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Women who were diagnosed as high-grade serous ovarian cancer
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2026-09-10 (Estimated); Study Completion 2027-09-10 (Estimated)

PRIMARY OUTCOMES:
Progression-Free-Survival | 36 months
  the length of time after surgical treatment for ovarian cancer that a patient lives without any signs or symptoms of the disease getting worse

CONTACTS AND LOCATIONS:
Overall Officials: Hongyu Xie, phD, Principal Investigator — Women's Hospital School Of Medicine Zhejiang University
Locations (1):
- Women's Hospital School of Medicine Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No